CLINICAL TRIAL: NCT06356064
Title: Investigation of The Effectiveness of Extracorporeal Shock Wave Therapy in Patients Diagnosed With Epin Calcanei: Comparison of Radial and Focus Applications
Brief Title: Radial or Focus Extracorporeal Shock Wave Therapy in Epin Calcanei
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2-23-3834
Record Dates: First submitted 2024-03-25; First posted 2024-04-10 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Spur, Heel
MeSH Terms: conditions — Heel Spur | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rESWT( Radial Extracorporeal shock wave therapy) (Experimental): rESWT(2.4 bar, 12 hz, 2000 beats), to painful calcaneal area, three sessions, once a week, for total of three weeks
  Interventions: Device: Extracorporeal shock wave therapy
- fESWT(Focused Extracorporeal shock wave therapy)) (Experimental): fESWT (0.14 bar, 14 hz, 1000 beats), to painful calcaneal area, three sessions, once a week, for total of three weeks
  Interventions: Device: Extracorporeal shock wave therapy

INTERVENTIONS:
Device: Extracorporeal shock wave therapy — Radİal ESWT and focus ESWT

SUMMARY:
Objective: The aim of the study was to investigate the effectiveness of radial and focused ESWT treatment on pain, function, and size of the calcaneal spur in patients with a clinical and radiological diagnosis of epin calcanei.

Methods: A total of 112 patients aged between 18 and 95 years were randomly divided into two groups: group 1 received rESWT (2.4 bar 12 hz 2000 beats), and group 2 received fESWT (0.14 bar 14 hz 1000 beats) three times a week for three weeks. All patients were evaluated using the Visual Analog Scale (VAS)-pain and Foot Function Index (FFI) before and after the treatment, at 4 weeks and 12 weeks. Epin size was measured radiographically in the patients before and after the treatment at the 12-week follow-up.

ELIGIBILITY:
Inclusion Criteria;

* Presence of heel pain for at least four weeks,
* Receiving no medical treatment, injection, physical or surgical treatment for the last four weeks and
* Agreed to participate in the study.

Exclusion Criteria:

* History of fracture or surgery,
* Polyneuropathy,
* Rheumatological diseases,
* Coagulation disorders,
* Tumor,
* Thrombosis,
* Soft tissue or bone infection,
* Pregnancy and lactation,
* Epilepsy,
* Presence of a pacemaker.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Before and after treatment baseline, 4th week, 12 th week
  0 min , 10 is maximum pain score
Functional Foot Index | Before and after treatment baseline, 4th week, 12 th week
  0 is no pain 10 is max pain, and 0 is no deficiency 10 is the maximum deficiency and 0 is no activity limitation 10 is the maximum activity limitation score.

SECONDARY OUTCOMES:
Radiographic assesment, epin size | Before and after treatment baseline, 4th week, 12 th week
  A decrease in the size of the epin is an indicator of recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Özge TEZEN, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
participant data will not share